CLINICAL TRIAL: NCT04142801
Title: Efficacy of the Memory Motivation (MEMO) Web Application for Cognitive and Behavioral Training in Patients With Neurocognitive Disorders
Brief Title: Efficacy of the Memory Motivation (MEMO) Web Application Training
Acronym: MeMo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Innovation Alzheimer (Other)
Collaborators: Alzheimer's Association (Other); Centre Hospitalier Universitaire de Nice (Other); Université de Nice Sophia Antipolis (Other)
Responsible Party: Principal Investigator, Philippe robert, MD, PhD, Professor of Psychiatry, Innovation Alzheimer
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-A00879-42
Record Dates: First submitted 2019-10-19; First posted 2019-10-29 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Neurocognitive Disorders
Keywords: Cognition; motivation; technology; non pharmacological intervention
MeSH Terms: conditions — Neurocognitive Disorders | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: regular use of a web application at home to train cognition and behavior
Who Masked: Participant, Investigator
Masking Description: Randomization for the allocation of the patient in each group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MeMo group (Experimental): MeMo group: experimental: regular use at home of the Memo web application In the Memo group patients were instructed on how to use the application, and allowed to train for 12 weeks. It was also explained that this training needed to be done regularly on a basis of 4 sessions of 30 minutes each per week.
  Interventions: Device: MeMo web application
- Control group (Placebo Comparator): Regular follow up at the memory center without cognitive training
  Interventions: Other: Control group

INTERVENTIONS:
Device: MeMo web application — The patient betwenn 2 consultation could use the application MeMo. MeMo is a web application that can thus be used on any web browser (computer or tablet). On tablet, the application can be installed on home screen to look like a native app, and used offline.
  Arms: MeMo group
Other: Control group — the patient have the classical follow up at the memory center (consultation)
  Arms: Control group

SUMMARY:
Memory, attentional, and behavioural symptoms are the clinical hallmarks of Neurocognitive disorders (NCD) such as Alzheimer's disease and related disorders. The World Health Organisation (WHO) guidelines for risk reduction of cognitive decline and dementia indicate that Cognitive training may be offered to older adults with normal cognition and with mild cognitive impairment to reduce the risk of cognitive decline and/or dementia. The use of Information and Communication Technologies (ICT) in the health domain is progressively expanding. The Alzheimer Innovation Association have developed MeMo (Memory Motivation) a free web application that can be used at home by patients.

The objective of the present study was to assess the effectiveness of employing the MeMo platform on cognitive performance in patients suffering from NCD.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the effectiveness of the MeMo cognitive training exercise platform in patients suffering from neurocognitive disorders. These exercises ,have been developed by the association Innovation Alzheimer and the CoBTeK research team, located with the Nice memory Center at the Institut Claude Pompidou. MeMo can be used freely at home by patients. More specifically, it is a randomized controlled study that aims to compare the evolution of activities cognition and behavior between patients not using these exercises, and patients using these exercises for 12 weeks, 4 sessions per week.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient consulting the Memory center
* older than 60 years old
* Mini Mental State examination score (MMSE) between 16 and 28 / 30
* met the DSM 5 diagnoses of mild neurocognitive disorders (mild NCD) or major neurocognitive disorders (Major NCD).

Exclusion Criteria:

* Patients not able to read and write French
* presence of a hearing or major visual impairment
* a history of premorbid mental retardation
* had already used the MeMo application
* were presently involved in structured memory training activities.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2019-02-02 (Actual); Study Completion 2019-08-10 (Actual)

PRIMARY OUTCOMES:
Change is being assessed with the Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE) | Base line, Week 12
  To score the IQCODE, add up the score for each question and divide by the number of questions. For the long IQCODE, divide by 26.

SECONDARY OUTCOMES:
Change in attention is is being assessed with the DSST | Base line, Week 12
  Digit Symbol Substitution Test (attentional task)
Change in frontal functioning is being assessed with the FAB | Base line, Week 12
  the Frontal Assessment Battery: Score 0 (healthy) - 18 (pathology)
Change in behavior is being assessed with the NPI | Base line, Week 12
  Neuropsychiatric Inventory score 0 (healthy) - 134 (pathology)
IA-C | Base line, Week 12
  Change in motivation is being assessed with theApathy inventory, clinician version score 0 (healthy)- 12 (pathology)

CONTACTS AND LOCATIONS:
Locations (1):
- CoBtek lab, Institut Claude Pompidou, Nice, France

REFERENCES:
- [Derived] Robert P, Manera V, Derreumaux A, Ferrandez Y Montesino M, Leone E, Fabre R, Bourgeois J. Efficacy of a Web App for Cognitive Training (MeMo) Regarding Cognitive and Behavioral Performance in People With Neurocognitive Disorders: Randomized Controlled Trial. J Med Internet Res. 2020 Mar 11;22(3):e17167. doi: 10.2196/17167. PMID 32159519